CLINICAL TRIAL: NCT00828295
Title: A Multicenter, Double-blind, Randomized, Parallel Group, Stratified Study to Assess the Safety and Efficacy of Single IV Doses of Palonosetron to Prevent Postoperative Nausea and Vomiting in Pediatric Patients
Brief Title: Safety and Efficacy of Palonosetron IV to Prevent Postoperative Nausea and Vomiting in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALO-07-29
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; palonosetron; pediatric
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 mcg/kg arm (Experimental): Single dose IV Palonosetron 1 mcg/kg (up to a maximum total dose of 0.075 mg)
  Interventions: Drug: palonosetron
- 3 mcg/kg arm (Experimental): Single dose IV Palonosetron 3 mcg/kg (up to a maximum total dose of 0.25 mg)
  Interventions: Drug: palonosetron

INTERVENTIONS:
Drug: palonosetron — palonosetron IV 1 mcg/kg
  Arms: 1 mcg/kg arm
Drug: palonosetron — palonosetron 3mcg/kg IV
  Arms: 3 mcg/kg arm

SUMMARY:
The objective of the study is to assess the safety and efficacy of two doses of IV palonosetron each administered as a single dose for the prevention of postoperative nausea and vomiting through 72 hours postoperatively in children aged 28 days up to 16 years inclusive undergoing surgical procedures requiring general endotracheal inhalation anesthesia.

ELIGIBILITY:
MAIN INCLUSION CRITERIA

* Male or female patient aged more than 28 days (full term) up to and including 16 years.
* Inpatient scheduled to undergo surgical procedures requiring general endotracheal anesthesia, including:

  * ear, nose and throat surgery;
  * eye surgery;
  * orchidopexy;
  * plastic reconstructive surgery;
  * herniorraphy;
  * orthopedic surgery).
* American Society of Anesthesiologists (ASA) physical status I, II or III.
* Patient scheduled to receive nitrous oxide during the maintenance phase of anesthesia.
* Patient scheduled to be hospitalized for at least 72 hours after wake up of surgery
* For female of childbearing potential: the patient and her parent(s)/legal guardian(s) were counseled on the importance of not becoming pregnant before or during the study and the patient must have a negative pregnancy test at the pre-treatment visit and at the study treatment visit.

MAIN EXCLUSION CRITERIA

* For infant aged more than 12 months: a history of gastro-esophageal reflux.
* For patient aged 28 days to 6 years: patient who received any investigational drugs within 90 days prior to Day 1. For patient aged 6 up to 16 years inclusive: patient who received any investigational drugs within 30 days prior to Day 1.
* Patient scheduled to undergo emergency surgery.
* Patient scheduled to receive regional (spinal) anesthesia in conjunction with general endotracheal anesthesia.
* Patient scheduled to receive propofol during the maintenance phase of anesthesia.
* Patient with vomiting from any organic cause.
* Any drug with a potential anti-emetic effect within 24 hours prior to the administration of anesthesia.
* Any vomiting, retching, or nausea in the 24 hours preceding the administration of anesthesia.

Ages: 28 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (5):
  - Federal State Institution Central Research Institute of Traumatology and Orthopedics n.a. N.N. Priorov under the Federal Agency for High-Tech Medical Care, Moscow
  - Federal State Institution Moscow Research Institute of Pediatrics and Pediatric Surgery under the Federal Agency for High-Tech Medical Care, Moscow
  - Federal State Institution St. Petersburg Research Institute of Ear, Throat, Nose and Speech under the Federal Agency for High-Tech Medical Care, Saint Petersburg
  - State Higher Educational Institution: "St. Petersburg State Pediatric Medical Academy under the Federal Agency for Healthcare and Social Development", Saint Petersburg
  - State Healthcare Institution 'Regional Pediatric Clinical Hospital', Yaroslavl
- Ukraine (8):
  - Cherkassy Regional Hospital, Pediatric Surgery Department, Cherkassy
  - Regional Children's Clinical Hospital. Dnipropetrovsk State Medical Academy, Pediatric Surgery Department, Dnipropetrovsk
  - M.Gorkyi Donetsk National Medical University, Pediatric Surgery Department; Children's Regional Clinical Hospital, Donetsk
  - Regional Children's Hospital, ENT Department, Ivano-Frankivsk State Medical University, ENT Department, Ivano-Frankivsk
  - Specialized Children's Hospital "OKHMATDYT", Orthopedics and Traumatology Department, O.O. Bohomolets National Medical University, Pediatric Surgery Department, Kyiv
  - Ukrainian Specialized Children's Hospital "OKHMATDYT", Anesthesiology and Intensive Care Department, P.L. Shupyk National Medical Academy of Postgraduate Education, Pediatric Anesthesiology and Intensive Care Department, Kyiv
  - Ukrainian Specialized Children's Hospital "OKHMATDYT", ENT Department, P.L. Shupyk National Medical Academy of Postgraduate Education, Pediatric ENT Department, Kyiv
  - Children's Clinical Hospital "OKHMATDYT", Institute of Congenital Pathology under the Academy of Medical Sciences of Ukraine, Lviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 19 August 2008. Last patient completed: 27 December 2008.
  A total of 12 Investigators from two countries (Russia and Ukraine) participated in the study. The study was conducted at 4 sites in Russia and 8 sites in Ukraine.
Period: Overall Study
Arm/Group | 1 mcg/kg Arm | 3 mcg/kg Arm
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mcg/kg Arm | 3 mcg/kg Arm | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Customized [Number; unit: participants]
  <2 years | 3 | 4 | 7
  2 to <6 years | 18 | 16 | 34
  6 to <12 years | 29 | 33 | 62
  12 to <17 years | 25 | 22 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 46 | 46 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 75 | 75 | 150
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ukraine | 48 | 49 | 97
  Russian Federation | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With no Emetic Episodes in the Overall Time Period 0-72 Hours Post-operatively
Time Frame: 0-72 hours post-operatively
Population: The Full Analysis Set (FAS) included all randomized patients, who received the study drug, had general anesthesia and surgery. Following the intent-to-treat principle, patients were assigned to the study treatment group according to the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1 mcg/kg Arm | 3 mcg/kg Arm
Number analyzed (Participants) | 75 | 75
percentage of patients | 88.0 [78.4 to 94.4] | 84.0 [73.7 to 91.4]

2. Secondary Outcome: Proportion of Patients With Complete Response 0-24 Hours
Description: Complete Response defined as no vomiting, no retching, and no use of rescue medication
Time Frame: 0-24 hours
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1 mcg/kg Arm | 3 mcg/kg Arm
Number analyzed (Participants) | 75 | 75
percentage of patients | 88.0 [78.4 to 94.4] | 84.0 [73.7 to 91.4]

ADVERSE EVENTS:
Time Frame: During the study, all adverse events were recorded and Patients stayed in the study for 22 days as a maximum. Duration of the safety follow up was 14 days after the patient completed the study for non Serious adverse events.
Description: Serious AEs were followed up until resolution/or reached a stable condition/or until subject lost to follow-up, Safety Set/SAF included all randomized patients assigned to treatment group according to actual treatment received. SAF had 74 and 76 patients/1 mcg/kg 3 mcg/kg group respectively/since one patient randomized 1 mcg/kg was treated 3 mcg/kg
Arm/Group | 1 mcg/kg Arm | 3 mcg/kg Arm
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 29/74 | 32/76
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mcg/kg Arm (N=74) | 3 mcg/kg Arm (N=76)
Procedural pain (Injury, poisoning and procedural complications) | 20 (20) | 19 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Asthenia (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (7)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No